CLINICAL TRIAL: NCT04996576
Title: Infrazygomatic Versus Intranasal Injection Approaches of Sphinopalatine Ganglion Blockade Effect on Surgical Field in Functional Endoscopic Sinus Surgeries
Brief Title: Infrazygomatic Versus Intranasal Injection Sphinopalatine Ganglion Blockade Effect on Surgical Field in FESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Wael Elswefi, principal investigator, Ain Shams University
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: sphinopalatine block in FESS
Record Dates: First submitted 2021-07-16; First posted 2021-08-09 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Nasal Polyps
MeSH Terms: conditions — Nasal Polyps

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intranasal injection approach sphinopalatine ganglion block (Active Comparator): Then in one nasal side (intranasal injection group) will be chosen randomly (right or left) by closed envelopes method 2 ml Lidocaine with Epinephrine 1/200000 will be injected posterior to meatus of middle concha to block terminal nerve branches of sphinopalatine ganglia and 2 ml saline will be injected in the same place in the other nasal side (to prevent surgeon expectation of intra nasal group by seeing injection site in one side only) by surgeon assistant who will be blind for the injection content.
  Interventions: Procedure: intranasal injection approach of sphinopalatine ganglion block
- infrazygomatic approach sphinopalatine ganglion block (Active Comparator): In the side saline only given by the intranasal injection A lateral fluoroscopic view of the face will be obtained with the C-arm by superimposing the mandibular rami on top of each other spinal needle with a slightly bent tip is inserted with lateral fluoroscopic guidance. superiorly and medially toward the sphinopalatine fossa.
  (AP) view intermittently obtained to check the depth 0.2 mL of contrast material will be injected to rule out intravascular spread and confirm spread of the dye within the sphinopalatine fossa .Local anesthetic, such as 2 mL of 1% lidocaine will be slowly injected
  Interventions: Procedure: infrazygomatic approach sphinopalatine ganglion block

INTERVENTIONS:
Procedure: infrazygomatic approach sphinopalatine ganglion block — A lateral fluoroscopic view of the face will be obtained with the C-arm by superimposing the mandibular rami on top of each other spinal needle with a slightly bent tip is inserted with lateral fluoroscopic guidance. superiorly and medially toward the sphinopalatine fossa.
  (AP) view intermittently obtained to check the depth 0.2 mL of contrast material will be injected to rule out intravascular spread and confirm spread of the dye within the sphinopalatine fossa .Local anesthetic, such as 2 mL of 1% lidocaine will be slowly injected
  Arms: infrazygomatic approach sphinopalatine ganglion block
Procedure: intranasal injection approach of sphinopalatine ganglion block — method 2 ml Lidocaine with Epinephrine 1/200000 will be injected posterior to meatus of middle concha to block terminal nerve branches of sphinopalatine ganglia
  Arms: intranasal injection approach sphinopalatine ganglion block

SUMMARY:
This study aimed to show the effect of sphinopalatine ganglion blockade on surgical field, hemodynamics and postoperative pain in FEES operation.

DETAILED DESCRIPTION:
Functional endoscopic sinus surgery (FESS) is a minimally invasive, effective surgical technique that is commonly used to treat chronic rhino sinusitis and nasal polyposis.

Intra-operative bleeding obscures the surgical view and increases the likelihood of iatrogenic complications. There are many factors that can affect the amount of bleeding experienced during surgery including both patient and surgical factors. These include severe forms of chronic sinusitis with nasal polyposis which is associated with increased vascularity, use of anticoagulant therapy, bleeding disorders, active infection, vascular tumor on the surgical site and revision surgery may affect bleeding on surgical site.

Sphenopalatine ganglion (SPG) is the main sensory innervation to the nasal mucosa.

The Sphenopalatine ganglion block (SPGB) is one of the regional anesthetic techniques that were used effectively before removal of nasal packing and in patients undergoing endoscopic sinus surgery under general anaesthesia to control bleeding or for postoperative analgesia

ELIGIBILITY:
Inclusion Criteria:

* Patients of ASA physical status I-II.

Exclusion Criteria:

* Patients of ASA physical status III or above.
* Patients with clinically significant cardiovascular, pulmonary or hepatic disease.
* Patients with bleeding diathesis or on anticoagulant therapy.
* Age less than 21 years.
* Mentally disabled patients.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
surgical field quality | during the surgery
  bloodless clear surgical field will be assessed for each side by surgeon using five categories categories.
  1. = uncontrolled bleeding.
  2. = severe bleeding, surgical conditions distorted immediately afterwards suctioning.
  3. = moderate bleeding, frequent suctioning required, visibility of the surgical field is moderate.
  4. = slight bleeding, occasional suctioning required, visibility of the surgical field is good.
  5. = no bleeding almost bloodless surgical field.

SECONDARY OUTCOMES:
blood pressure | during the surgery and after the surgery( up to 24 hours)
  Intraoperative blood pressure changes will be observed every 10 minutes and will be compared between the two sides in the unit mmHg Postoperatively, patients will be observed in the postanesthesia care unit (PACU). During the observation period, arterial blood pressure will be continuously monitored every 15 minutes for 1 hour. Patients meeting PACU discharge criteria will be transferred to the surgical ward. blood pressure will be reported every 4 hours for 24 hours.
heart rate | during the surgery and after the surgery( up to 24 hours)
  intraoperative heart rate will be compared between the two sides in the unit beat per minute Postoperatively, patients will be observed in the postanesthesia care unit (PACU). During the observation period, heart rate will be continuously monitored every 15 minutes for 1 hour. Patients meeting PACU discharge criteria will be transferred to the surgical ward. heart rate will be reported every 4 hours for 24 hours
Postoperative pain | immediately after the surgery and 12 , 24 hours after the surgery
  Postoperative pain will be assessed and patient will be asked to compare between the two nasal sides, in the PACU and at 6, 12 and 24 hours after surgery with a 10-cm visual analog scale (VAS) (0 = no pain, 10 = most severe pain). Pain severity will be divided into 3 groups: mild, score of <4; moderate, score of 4 to 6; and severe >6
postoperative epistaxis | after the surgery( up to 24 hours)
  epistaxis
postoperative infection | after the surgery( up to 24 hours)
  nasal infection

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Ain shams university hospitals, Cairo
  - Ain Shams university, Cairo